CLINICAL TRIAL: NCT02344498
Title: Treatment of Hepatitis B in Resource-limited Settings - a Pilot Program in East Africa
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Addis Ababa University (Other); The Research Council of Norway (Other); University of Agder (Other); South-Eastern Norway Regional Health Authority, Norway (Unknown); St. Paul's Hospital Millennium Medical College, Ethiopia (Other); Haramaya University,Ethiopia (Unknown)
Responsible Party: Principal Investigator, Asgeir Johannessen, Researcher / project manager, Oslo University Hospital
Other Study IDs: 2014/1146
Record Dates: First submitted 2015-01-16; First posted 2015-01-26 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Hepatitis B
Keywords: Liver cirrhosis; Antiviral agents; Liver diseases
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis; Liver Diseases | interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Urban: HBV patients in Addis Abeba. Eligible patients treated with tenofovir disoproxil fumarate 245 mg OD.
  Interventions: Drug: Tenofovir disoproxil
- Rural: HBV patients in Adama, Afar, Jigjiga and Jimma. Eligible patients treated with tenofovir disoproxil fumarate 245 mg OD.
  Interventions: Drug: Tenofovir disoproxil

INTERVENTIONS:
Drug: Tenofovir disoproxil

SUMMARY:
Viral hepatitis kills nearly one million people each year, even though effective treatment exists. The aim of this study is to establish a treatment protocol for hepatitis B, which is simple and cheap enough to be implemented in resource-limited settings.

DETAILED DESCRIPTION:
Chronic viral hepatitis is a major health problem globally. Each year nearly one million deaths are attributable to either hepatitis B or C. In Ethiopia 5-10% of the general population are infected with hepatitis B. Oral antiviral treatment of hepatitis B exists, but high costs and advanced laboratory requirements have been barriers to offer such treatment in resource-limited settings, resembling the situation in treatment of HIV/AIDS a decade ago.

The present study will investigate a simplified approach to hepatitis B treatment in resource-limited settings, inspired by the recent success of HIV treatment in such settings. The critical research question is how to identify patients with expected benefit of treatment in the absence of advanced laboratory support. A WHO expert panel recently suggested treatment criteria for use in settings without advanced laboratory facilities, but these criteria have not yet been tested out in real life. The present study will build on and develop the WHO approach to treatment of hepatitis B, aiming to develop a treatment protocol that can be feasible in other resource-limited countries. The potential public health benefit for poor people in low- and middle-income countries is substantial.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults (≥18 years) residing in Ethiopia who are HBsAg positive

Exclusion Criteria:

* Children <18 years, other terminal disease (cancer etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults with a positive HBsAg rapid test are eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 7350 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Death, HCC or decompensated cirrhosis | 3 years
  Patients will be reviewed every 3-6 months with liver function tests and/or ultrasound to detect the proportion of participants who develop liver decompensation or hepatocellular carcinoma.

SECONDARY OUTCOMES:
Viral suppression and genotypic resistance | 3 years
  Proportion of patients with viral load suppression and absence of resistance after >1 year of antiviral treatment.
Regression of liver inflammation/fibrosis | 3 years
  Proportion of patients with normalization of ALT and improvement of liver stiffness (by transient elastography)
Adherence to therapy | 3 years
  Proportion of patients with >95% adherence measured by pill count and visual analogue scale

OTHER OUTCOMES:
Sensitivity and specificity of HBsAg rapid tests | 1 year
  Sensitivity and specificity of commonly used HBsAg rapid tests compared to a gold standard ELISA method

CONTACTS AND LOCATIONS:
Overall Officials: Asgeir Johannessen, MD PhD, Principal Investigator — Oslo University Hospital; Nega Berhe, MD PhD, Principal Investigator — Addis Abeba University
Locations (1):
- St Paul Hospital Millennium Medical College, Addis Ababa, Addis Abeba, Ethiopia

REFERENCES:
- [Derived] Rossvoll L, Desalegn H, Gudissa FG, Birhanu D, Hussen A, Cheneke W, Jeylan A, Debela EA, Yusuf M, Sugule A, Berhanu N, Gudina EK, Orlien SM, Stockdale AJ, Berhe N, Johannessen A. Treatment of chronic hepatitis B in Ethiopia: 1-year results from a real-life, multicentre, prospective cohort study. Lancet Glob Health. 2025 Nov;13(11):e1914-e1923. doi: 10.1016/S2214-109X(25)00309-2. PMID 41109262
- [Derived] Desalegn H, Orlien SMS, Aberra H, Mamo E, Grude S, Hommersand K, Berhe N, Gundersen SG, Johannessen A. Five-year results of a treatment program for chronic hepatitis B in Ethiopia. BMC Med. 2023 Sep 29;21(1):373. doi: 10.1186/s12916-023-03082-4. PMID 37775742
- [Derived] Desalegn H, Aberra H, Berhe N, Medhin G, Mekasha B, Gundersen SG, Johannessen A. Predictors of mortality in patients under treatment for chronic hepatitis B in Ethiopia: a prospective cohort study. BMC Gastroenterol. 2019 May 15;19(1):74. doi: 10.1186/s12876-019-0993-1. PMID 31092203
- [Derived] Aberra H, Desalegn H, Berhe N, Mekasha B, Medhin G, Gundersen SG, Johannessen A. The WHO guidelines for chronic hepatitis B fail to detect half of the patients in need of treatment in Ethiopia. J Hepatol. 2019 Jun;70(6):1065-1071. doi: 10.1016/j.jhep.2019.01.037. Epub 2019 Mar 28. PMID 30929749
- [Derived] Desalegn H, Aberra H, Berhe N, Mekasha B, Stene-Johansen K, Krarup H, Pereira AP, Gundersen SG, Johannessen A. Treatment of chronic hepatitis B in sub-Saharan Africa: 1-year results of a pilot program in Ethiopia. BMC Med. 2018 Dec 17;16(1):234. doi: 10.1186/s12916-018-1229-x. PMID 30554571
- [Derived] Aberra H, Gordien E, Desalegn H, Berhe N, Medhin G, Mekasha B, Gundersen SG, Gerber A, Stene-Johansen K, Overbo J, Johannessen A. Hepatitis delta virus infection in a large cohort of chronic hepatitis B patients in Ethiopia. Liver Int. 2018 Jun;38(6):1000-1009. doi: 10.1111/liv.13607. Epub 2017 Oct 20. PMID 28980394
- [Derived] Aberra H, Desalegn H, Berhe N, Medhin G, Stene-Johansen K, Gundersen SG, Johannessen A. Early experiences from one of the first treatment programs for chronic hepatitis B in sub-Saharan Africa. BMC Infect Dis. 2017 Jun 19;17(1):438. doi: 10.1186/s12879-017-2549-8. PMID 28629395
- [Derived] Desalegn H, Aberra H, Berhe N, Gundersen SG, Johannessen A. Are non-invasive fibrosis markers for chronic hepatitis B reliable in sub-Saharan Africa? Liver Int. 2017 Oct;37(10):1461-1467. doi: 10.1111/liv.13393. Epub 2017 Mar 23. PMID 28222249